CLINICAL TRIAL: NCT05944445
Title: The Incidence of Linezolid-induced Thrombocytopenia (LIT) in Critically Ill Patients, the Risk Factors for LIT and Time to Events (LIT, Recovery)
Brief Title: The Incidence of Linezolid-induced Thrombocytopenia (LIT) in Critically Ill Patients, the Risk Factors for LIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed Abdeltawab, Clinical pharmacist, Helwan University
Other Study IDs: 11041989
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Thrombocytopenia; Drugs
Keywords: Linezolid; Thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Linezolid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm group: Adult critically ill patients admitted to ICU for different indications
  Interventions: Drug: Linezolid 600 mg

INTERVENTIONS:
Drug: Linezolid 600 mg — Linezolid 600mg injection

SUMMARY:
* To identify the incidence of LIT among critically ill patients, as limited studies have only addressed this population.
* To evaluate the impact of several factors on the incidence of LIT, the time to onset of LIT, and the time to recovery of platelets.
* To study the effect of concurrent medications (enoxaparin, unfractinated heparin, piperacillin, carbapenems, tigecycline, fluconazole or voriconazole, digoxin, amiodarone, acetaminophen, tirofiban, statins, and antiepileptics) frequently used in critically ill patients on the incidence of LIT.
* To investigate the impact of possible medications with an antioxidant effect on the prevention of LIT.
* To assess the impact of LIT on composite end point (mortality, bleeding, and length of stay)

ELIGIBILITY:
Inclusion Criteria:

* All adult patients, age > or = 18 years old, admitted to the ICU with different indications.
* candidates for intravenous linezolid therapy for > or =1 day.

Exclusion Criteria:

* Taking any myelosuppressive drug.
* Baseline platelets < 50000.
* Patients with hematological malignancy.
* COVID-19 patients.
* Patients with immune thrombocytopenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted to ICU for different indications
Sampling Method: Non-Probability Sample
Enrollment: 310 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Linezolid-induced thrombocytopenia (LIT) thrombocytopenia | One year
  Defined as platelets < 150000 OR decrease > 50% of baseline platelets.

SECONDARY OUTCOMES:
Time to the onset of LIT | One year
  Defined as platelets < 150000 OR decrease > or = 50% of baseline platelets.
time to platelet recovery | One year
  after having thrombocytopenia, regardless of discontinuation of linezolid, recovery is defined as the restoration and maintenance of platelet counts > 70% of baseline values
Incidence of clinical outcomes | One year
  Incidence of clinical outcomes (bleeding, mortality, length of stay, need for platelet or blood transfusion).

CONTACTS AND LOCATIONS:
Overall Officials: Abdelhameed I Ebid, Study Director — Helwan University, faculty of pharmacy; Mahmoud I Mostafa, Study Director — Helwan University, faculty of pharmacy
Locations (1):
- 15 May hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided